CLINICAL TRIAL: NCT03701425
Title: Impact of Interventions With a Diet and Exercise on the Cardio-metabolic Status in Multi-risk Population
Acronym: PANDEMONIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Juan Antonio Suárez Cuenca, Ph D, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 083.2018
Record Dates: First submitted 2018-07-12; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome x; Mediterranean Diet
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Masking Description: Random assignment, through software, to 4 treatment groups: one, first consume the Mediterranean and exercise plan, second group will be given only nutritional plan with Mediterranean diet, the third group only exercise plan, and the fourth control group which will give a low standard low fat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mediterranean diet and exercise plan (Experimental): Random assignment, through software, to 4 groups of treatment: consume the Mediterranean diet: according to the definition, with the distribution of macronutrients: Protein contribution 0.8-1.2 gram, Carbon Hydrates 45-50% Lipids 30% An exercise plan: The "classic" exercise program who they will carry out a 5-minute warm-up program with active mobilizations. After that, they will perform intervals of 5 min with resistance to maintain the heart rate prescribed, with active breaks of 1 - 2 min, 4 repetitions. At the end, there will be a return to calm The program of high-intensity anaerobic exercise will consist of a 5-minute warm-up , followed by 5 sets of isokinetic exercise with protocol "November 20", rest of 90 s between series. The program will be done 3 times per week for 12 weeks.
  Interventions: Dietary Supplement: Mediterranean diet and exercise plan
- Mediterranean diet (Experimental): Random assignment, through software, to 4 groups of treatment: consume the Mediterranean diet: according to the definition, with the following distribution of macro nutrients: Protein contribution 0.8-1.2 gram Carbon Hydrates 45-50% Lipids 30%
  Interventions: Dietary Supplement: Mediterranean diet and exercise plan
- Only exercise (Active Comparator): An exercise plan: The "classic" exercise program who they will carry out a 5-minute warm-up program with active mobilizations. After that, they will perform intervals of 5 min with resistance to maintain the heart rate prescribed, with active breaks of 1 - 2 min, 4 repetitions. At the end, there will be a return to calm The program of high-intensity anaerobic exercise will consist of a 5-minute warm-up , followed by 5 sets of isokinetic exercise with protocol "November 20", rest of 90 s between series. The program will be done 3 times per week for 12 weeks.
  Interventions: Dietary Supplement: Mediterranean diet and exercise plan
- Low standard low fat diet (Active Comparator): Random assignment, through software, to 4 groups of treatment: consume the low standard low fat diet: according to the definition, with the following distribution of macro nutrients:Protein contribution 0.8-1.2 Carbon Hydrates 45-50% Lipids 20%
  Interventions: Dietary Supplement: Mediterranean diet and exercise plan

INTERVENTIONS:
Dietary Supplement: Mediterranean diet and exercise plan — Mediterranean diet:
  Diet: according to the definition, with the following distribution of macro nutrients:
  Protein contribution 0.8-1.2 Carbon Hydrates 45-50% Lipids 30%

SUMMARY:
The diseases derived from Metabolic Syndrome caused 75% of the total deaths. It is more profitable to invest in prevention than in the treatment of most cardiovascular diseases. Several institutions consider prevention as one of the main priorities in public health.

Patients with Metabolic Syndrome, undergoing Mediterranean diet and exercise program, will have lower fat mass, greater lean mass and muscle strength; in addition to the lower expression of proinflammatory biomarkers, compared to those subjected to standard diet and exercise.

OBJECTIVE: To evaluate the changes in body composition and cardiovascular risk in the population with metabolic syndrome undergoing a Mediterranean diet program and / or controlled physical activity.

Design: Experimental, longitudinal design, controlled clinical trial, randomized. Population with Metabolic Syndrome in which the effect of Mediterranean diet and / or controlled physical activity will be compared on anthropometric parameters, body composition, cardiometabolic risk and plasma biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of metabolic syndrome.
* Patients diagnosed with overweight.
* Patients diagnosed with obesity.
* Patients with a diagnosis of systemic arterial hypertension.
* Patients diagnosed with type 2 diabetes mellitus.
* Patients with dyslipidemia.

Exclusion Criteria:

* Recent myocardial infarction
* Pregnancy
* Lactation
* In pharmacological treatment for weight loss.
* Cancer.
* Chronic kidney disease
* Liver failure
* Heart failure.
* Chronic obstructive pulmonary disease
* Depression
* Malabsorption syndrome
* Chronic diarrhea

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-12 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure the profiles of body composition in the different groups. | 3 months
  Measure the basal profiles of body composition (weight in kilograms and height in meters, body mass index in kg/m^2, bio impedance will be done by bioimpedance multifrequency, 8 points) in the different groups
Measure the profiles of pro inflammatory biomarkers. | 3 months
  Determine the basal pro-inflammatory biomarkers (interleukins 1 beta in picograms per liter , interleukin 2 in picograms per liter , interleukins 10 in picograms per liter ) in the 4 different groups.
Compare the profiles of body composition and proinflammatory biomarkers after the follow-up between the different groups in patients with metabolic syndrome. | 3 months
  To compare the profiles of body composition and proinflammatory biomarkers after a program of physical activity and feeding plan, in the different groups of patients with metabolic syndrome after the follow-up and classify by groups, responds or not responds for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Center "20 de Noviembre", ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No